CLINICAL TRIAL: NCT01829776
Title: Pilot Study on the Effect of the Free From Falls Program on Falls in People With Multiple Sclerosis
Brief Title: Pilot Study of Free From Falls Program in Multiple Sclerosis
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michelle Cameron, Neurologist, Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9257
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis
Keywords: Accidental falls; Multiple Sclerosis; Education; Exercise; Postural balance
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- education (Experimental): Educational intervention
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — This is an 8-week comprehensive fall prevention exercise and education program, with one 2-hour session each week, for people with MS, adapted from a similar program for older adults.

SUMMARY:
This pilot study will compare how often people with multiple sclerosis (MS) fall before participating in the Free From Falls (FFF) educational program, during the program, and for 8 weeks after the program. The protocol will also evaluate the accuracy, efficiency and convenience of an email survey to count how often people fall.

DETAILED DESCRIPTION:
This pilot study will recruit people with MS who report falling at least twice in the previous 2 months to participate in the FFF program. All subjects will record their falls and injurious falls on a daily basis for at least 3 weeks before the program, during the program and for 8 weeks after the program. The program will consist of a weekly 2 hour session. One hour of the session will be educational and one hour of the program will involve exercise. The outcome of this study will be change in fall rate between the periods before, during and after the program.

ELIGIBILITY:
Inclusion Criteria:

* MS of any type
* Age 18 years or older
* Able to walk at least 100 meters with intermittent or unilateral constant assistance (cane, crutch or braces) with or without resting
* Self-reported history of 2 or more falls in the previous 2 months
* Clinically stable MS with no relapses within 30 days
* Willing to provide informed consent
* Fluent in written and spoken English.
* Daily access to email and willing to respond to a daily email questionnaire

Exclusion Criteria:

* Serious psychiatric or medical conditions that would preclude reliable participation in the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in fall frequency per month (30 days) | difference between the wait period before the 8 week FFF program and the 8 weeks after the end of the 8 week FFF program
  The change in fall frequency between the wait period before the FFF program begins and 8 weeks after the program has ended.

SECONDARY OUTCOMES:
Relationship between paper and electronic fall calendars | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle H Cameron, MD, PT, Principal Investigator — Oregon Health & Science University, Portland VA Medical Center
Locations (1):
- Oregon Health and Science University and Portland VA Medical Center, Portland, Oregon, United States